CLINICAL TRIAL: NCT00236366
Title: Randomised, Double-Blind, Placebo-Controlled, Parallel-Group, Multicentre Trial To Investigate Durogesic™ In Comparison To Placebo In Subjects With Moderate To Severe Pain Induced By Osteoarthritis Of The Hip Or The Knee, Who Are In Need Of And Waiting For Hip Or Knee Replacement.
Brief Title: A Study of the Effect on Pain Control of Treatment With Fentanyl, Administered Through the Skin, Compared With Placebo in Patients With Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003004
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-12

CONDITIONS: Osteoarthritis; Arthritis
Keywords: Fentanyl; opioid analgesics; osteoarthritis; arthritis; transdermal administration
MeSH Terms: conditions — Osteoarthritis; Arthritis | interventions — Fentanyl

INTERVENTIONS:
Drug: fentanyl

SUMMARY:
The purpose of the study is to determine if fentanyl, delivered through the skin via an adhesive patch, has a superior pain-relieving effect compared with placebo in patients with osteoarthritis pain that is inadequately controlled by therapeutic treatment with weak opioids, which are often taken in combination with non-opioid analgesics.

DETAILED DESCRIPTION:
Chronic, non-cancer pain may result from injury or illness, such as osteoarthritis or rheumatoid arthritis, which causes suffering and a reduction in the quality of life. Opioids, such as fentanyl, are beneficial as potent pain-relieving drugs in patients with continuous pain. This is double-blind, parallel-group, placebo-controlled study to compare pain relief, and the effect on safety, functionality, and quality of life during treatment with fentanyl administered through the skin via adhesive patches ("transdermal system") with therapy with placebo in patients with osteoarthritis (OA). Specifically, patients with moderate to severe pain induced by osteoarthritis and for whom treatment with traditional pain medication (according to the World Health Organization [WHO] pain ladder, up to and including weak opioids) has failed to provide adequate pain relief, are eligible to enroll. After screening, patients enter a 1-week Run-In period, in which prior treatment with weak opioids, with or without non-opioid pain medication, continues. After this period, patients with moderate to severe pain are randomized to the fentanyl adhesive patch or placebo during the Double-Blind (Treatment) phase for 6 weeks. All patients, including those who discontinue or withdraw from the study, enter the Tapering-Off period, during which the medication is reduced gradually. Assessments of effectiveness include: Pain relief, determined with a Visual Analogue Scale (VAS) by means of an electronic pain diary updated by the patient at least twice daily; functionality, assessed by the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index; and quality of life, measured by the SF-36 Quality of Life Questionnaire. Safety assessments include identification of possible withdrawal symptoms at the end of the Tapering-Off period, measurement of vital signs at stated intervals, and incidence of adverse events throughout the study. The study hypothesis is that patients with osteoarthritis of the hip or knee whose pain is not adequately controlled by other pain-relieving medications will show an improvement in pain control after treatment with the fentanyl transdermal system. Fentanyl patches to deliver 25 micrograms/hour to 100 micrograms/hour, changed every 3 days, for 6 weeks; doses may be adjusted for adequate pain control; anti-nausea tablets (Metoclopramide, 10 milligrams[mg], and paracetamol tablets (500 mg; maximum 4 grams/day) as supplementary pain control

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis (OA) of the hip or the knee (as defined by the American College of Rheumatology) and radiological evidence of OA from the target joint
* patients must be in need of and waiting for hip or knee replacement
* patients with chronic pain for longer than 3 months for >=20 days/month
* patients with moderate to severe OA pain of the target joint (VAS score >=50 on a scale of 0-100), whose pain was not adequately controlled with weak opioids, with or without non-opioid pain medication
* women must be postmenopausal or using adequate contraception, have a negative pregnancy test at study initiation, and not be breastfeeding.

Exclusion Criteria:

* Patients who had previously failed fentanyl therapy or had discontinued treatment due to adverse events
* known allergy or hypersensitivity to fentanyl or to the adhesives
* patients being treated for depression or epilepsy
* patients who received sedative hypnotics, anaesthetics and/or muscle relaxants in the week preceding the Run-In Period
* patients experiencing another type of continuous pain that stands out in comparison with OA pain
* patients with major trauma to the target joints, infection in these joints, or irreversible damage to these joints during the 6 months before the study.

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2002-06; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Average Area Under the Curve Minus Baseline (AAUCMB) of pain relief, as measured by Visual Analogue Scale (VAS) scores for daily pain during the treatment period (6 weeks)

SECONDARY OUTCOMES:
SF-36 Quality of Life Questionnaire (QoL) and WOMAC questionnaire on Days 1 and 43 and at end of tapering-off period; adverse events throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.

REFERENCES:
- See also: Randomized, double-blind, placebo-controlled, parallel-group, multicentre trial to investigate DurogesicTM in subjects with moderate to severe pain induced by osteoarthritis of the hip or the knee. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=380&filename=CR003004_CSR.pdf